CLINICAL TRIAL: NCT04416789
Title: A Feasibility Study to Determine the Acceptability and Impact of an Exercise Intervention for Children With Neurodevelopmental Difficulties and Sleep Problems
Brief Title: Exercise Intervention for Sleep in Neurodevelopmental Disorders
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 237572
Record Dates: First submitted 2019-02-15; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2019-02

CONDITIONS: Neurodevelopmental Disorders; Sleep Disorder
Keywords: children; sleep; exercise; neurodevelopment; feasibility
MeSH Terms: conditions — Neurodevelopmental Disorders; Sleep Wake Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise programme — 1 session of trampolining/dry sports (1.5 hours) and 1 session of supervised swimming (1.5 hours) per week for 10 weeks.

SUMMARY:
There is a long-standing assumption that physical activity is an effective, non-pharmacological approach to improving sleep quality and quantity. However, objective and reliable data on this relationship are scarce for children with developmental disabilities.

Parent burnout in this population is high and there are many barriers to engagement with such interventions. This study aims to understand the feasibility of providing an exercise intervention for this population, and gathering parental views on the impact of such an intervention.

Depending on the outcome of this feasibilty study, larger scale interventions may be planned to further examine the impact of such an intervention.

DETAILED DESCRIPTION:
Exercise in this population:

The impact of exercise on sleep in children with developmental disabilities is so far tentative. Small-scale studies suggest increasing physical activity in children with neurodevelopmental disorders leads to increased sleep quality.

Recommendations from previous research have included that future studies should assess the benefit of a longer intervention period, and impact on the wider family. Our study design aims to address these two factors.

Method:

Feasibility study using a one sample pre-post design.

Recruitment:

Participants will be informed of the study during the standard clinic assessment run by the Community Paediatricians (Community Sleep Clinic Lambeth and Southwark). A "consent to be contacted" letter will be used to facilitate agreement for the research team to contact families to discuss the study in more detail. Families will then be contacted by a member of the team not directly linked to their care. Information will be given over the phone and the family invited to a study information session at which the study will be explained further, questions answered, and consent taken for those who wish to take part.

During and after completion of the intervention all participants will continue through the usual treatment pathway.

Figure one: participant flow diagram:

Baseline assessment - parent to complete 2 weeks of sleep diaries for child prior to intervention; child height and weight measurement.

Intervention - 1 session of swimming (1.5 hours) and 1 session of trampolining and dry sports (1.5 hours) per week for 10 weeks, totalling 20 x 1.5 hours. The intervention will be tailored to the level of ability for each participant (i.e. each exercise will have different levels of complexity). Details of the specifics of the intervention that will be undertaken by the participants is as above. The intervention will be provided by the 'London PE and Schools Sport Network'. This company is a well-known sports company in South London that specialise in providing sports coaching for children with additional needs.

End of intervention assessment - parent to complete 2 weeks of sleep diaries for child for last 2 weeks of intervention, and to complete Likert-scale and free-text questionnaires as below.

Definition of end of trial:

The trial will end 3 months after the last exercise session, when height and weight are recorded as the final measure at a face-to-face clinic appointment.

Sample:

This number is limited to the number of children the instructor can teach during a course of the intervention. The instructor has advised he can teach a maximum of 15 students. Data on age, gender, ethnicity, weight and medical diagnosis will be recorded

Outcome measures:

1. Acceptability of the intervention with respect to accessibility, journey to venue, appropriateness, likelihood to recommend to others
2. Attrition rate
3. Sleep diaries will be completed by parents/carers specifically to assess:

   * Bedtime
   * Time fell asleep (to then work out sleep latency/time to fall asleep)
   * Number of night wakings
   * Morning wake-up time
   * Estimated total sleep time per night for 2-weeks pre-intervention, and during the last 2 weeks of intervention for comparison
4. Parent reported effects on wellbeing of child and family scored on Likert Scale (see Parent-reported outcome measures, Appendix 1)
5. Measurement of Body Mass Index pre-intervention and at 3-months post-intervention at face-to-face clinic appointment

Study Timetable:

Month 1: Recruitment Month 2-4: Intervention, 2 sessions weekly for 10 weeks Month 5-7: Data collection Month 7-9: Data Analysis Month 10-12: Writing up

Eligibility Inclusion criteria

1. Diagnosed neurodevelopmental disability
2. Open to the Lambeth and Southwark Community Sleep Clinic
3. Age range: 5 years 0 months - 15 years 11months. Exclusion criteria

1) High risk safeguarding concerns 2) Health issues where the intervention has the potential to have an adverse effect on the child e.g. undiagnosed/untreated epilepsy

Criteria and procedures for subject withdrawal or discontinuation.

1. Injury or illness (physical or mental) that prevents the participant engaging in the activity.
2. Parental choice to remove participant from activity

ELIGIBILITY:
Inclusion Criteria:

Diagnosed neurodevelopmental disability Open to the Lambeth and Southwark Community Sleep Clinic Age range: 5 years 0 months - 15 years 11months.

Exclusion Criteria:

1. High risk safeguarding concerns
2. Health issues where the intervention has the potential to have an adverse effect on the child e.g. undiagnosed/untreated epilepsy

Ages: 5 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Children aged 5 years to 15 years 11 months attending the Community Sleep Clinic (a dedicated Sleep Clinic for children with neurodevelopmental disorders); all levels of disability will be catered for within the exercise intervention
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Acceptability of the exercise intervention to families | Collected in three months following end of intervention
  Measured by attrition rate
Acceptability of the exercise intervention to families | Collected in three months following end of intervention
  Measure by semi-structured questionnaire; how likely would you be to recommend the activity; how accessible was the venue; how appropriate was the activity to your child's needs; any other comments; with 5-point Likert scale

SECONDARY OUTCOMES:
Impact on the sleep pattern of partaking children | For 2 weeks prior to intervention, and for last 2 weeks of intervention
  Through sleep diary reporting (bedtime, time fell asleep, number of times woke in night, time of morning waking, estimated total sleep in hours)
Impact on the child and family's wellbeing | Collected within three months following end of intervention
  Through Likert scale reporting by parent for perceived impact on sleep pattern, general wellbeing, mood and behaviour, wellbeing of parent and/or family (made a lot worse, made a bit worse, no change, improved a bit, improved a lot, improved a great deal)

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Supporting data can be made available on request by contacting study lead